CLINICAL TRIAL: NCT01327807
Title: Cure Cystinosis International Registry
Acronym: CCIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cystinosis Research Foundation (Other)
Responsible Party: Principal Investigator, Jerry A. Schneider, Professor Emeritus of Pediatrics, Cystinosis Research Foundation
Other Study IDs: CCIR100913
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Cystinosis; Nephropathic Cystinosis; Renal Fanconi Syndrome
Keywords: Registries; Cystinosis; Nephropathic Cystinosis; Renal Fanconi Syndrome; Cystine; Kidney; Rare Diseases
MeSH Terms: conditions — Cystinosis; Fanconi Syndrome; Rare Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cystinsosis patients: Those with a diagnosis of cystinosis.

SUMMARY:
Cure Cystinosis International Registry (CCIR) is an online, patient self-identifying registry developed by medical and scientific experts specifically for the cystinosis community.

CCIR's sole purpose is to identify people with cystinosis worldwide in an effort to accelerate novel treatments and a cure for cystinosis.

CCIR provides a safe and secure platform for:

* sharing anonymous medical information about cystinosis with researchers, clinicians and patients
* disseminating information about research opportunities
* connecting researchers/investigators and prospective participants *

Interested cystinosis patients may register themselves with CCIR online at http://www.cystinosisregistry.org.

* No personal information is shared outside of CCIR. Individual identities are known only to appropriate CCIR staff. If a participant is matched to a clinical trial, the participant receives a notice from CCIR, after which they can decide whether they wish to contact the study sponsor.

DETAILED DESCRIPTION:
Significance and Purpose:

Many different resources and tools are necessary to make significant advances in medical research. Progress in rare diseases such as cystinosis can often be impeded by the lack of information available about the disease and limited access to volunteers eligible for clinical trials. Therefore, patients who are willing to provide information about how the disease has affected them and also make themselves available to participate in trials are among the most valuable resources the investigators have to fight a disease. However, the research community desperately needs the right tool that will permit access to these resources.

A tool widely used to conveniently collect both data about a disease and information about potential clinical trial participants is a patient registry. A patient registry is any system that allows for the organized collection of data about disease outcomes in affected populations for a scientific, clinical, or policy purpose. The Cystinosis Research Foundation (CRF) has aligned itself with cystinosis medical experts and organizations worldwide to create the first ever international, online patient registry for cystinosis, Cure Cystinosis International Registry (CCIR). The express purpose of CCIR is to make anonymous information available to the research community and thus promote accelerated research in advanced treatments and ultimately a cure for cystinosis.

Objectives:

The objectives of CCIR are:

* Evaluate epidemiology and clinical characteristics of cystinosis around the world.
* Evaluate and compare the diagnosis, treatment, and kidney transplant rates among cystinosis communities from different geographical areas.
* Enhance the understanding of how cystinosis affects quality of life.

CCIR Registration:

Interested cystinosis patients may register themselves with CCIR online at http://www.cystinosisregistry.org. Registration is easy and secure. Simply go to the website and create a CCIR account and complete a survey. The CCIR website is currently available in English and Spanish, and will soon be available in French, Portuguese, and possibly other languages.

Benefits to CCIR participants include instant access to the registry's accumulated survey results (reported as anonymous group data), and opportunities to submit questions to cystinosis experts and to learn of clinical trial opportunities. No personal information is shared outside of CCIR. Individual identities are known only to appropriate CCIR staff.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystinosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: International cystinosis community
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2010-08; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Age at treatment initiation and the effect on disease outcomes | Lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Schneider, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Result] Cherqui S. Cysteamine therapy: a treatment for cystinosis, not a cure. Kidney Int. 2012 Jan;81(2):127-9. doi: 10.1038/ki.2011.301. PMID 22205430
- [Result] Gangoiti JA, Fidler M, Cabrera BL, Schneider JA, Barshop BA, Dohil R. Pharmacokinetics of enteric-coated cysteamine bitartrate in healthy adults: a pilot study. Br J Clin Pharmacol. 2010 Sep;70(3):376-82. doi: 10.1111/j.1365-2125.2010.03721.x. PMID 20716238